CLINICAL TRIAL: NCT06425159
Title: A Phase 2/3 Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of BHV-7000 as Adjunctive Therapy in Subjects With Idiopathic Generalized Epilepsy With Generalized Tonic-clonic Seizures, With Open-label Extension
Brief Title: A Study to Determine if BHV-7000 is Effective and Safe in Adults With Idiopathic Generalized Epilepsy With Generalized Tonic-clonic Seizures
Acronym: SHINE
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV7000-304; 2023-508812-45-00 (Other: EU CTR)
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Generalized Epilepsy
Keywords: Idiopathic Generalized Epilepsy; Generalized; Epilepsy; tonic-clonic; generalized tonic-clonic; tonic; clonic; seizure; refractory epilepsy; generalized tonic-clonic alone; juvenile myoclonic epilepsy; juvenile absence epilepsy
MeSH Terms: conditions — Epilepsy, Generalized; Epilepsy, Idiopathic Generalized; Epilepsy; Seizures; Drug Resistant Epilepsy; Myoclonic Epilepsy, Juvenile; Epilepsy, Absence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV-7000 75 mg (Active Comparator)
  Interventions: Drug: BHV-7000
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-7000 — BHV-7000 75mg. Participants will take blinded investigational product (IP) once daily
  Arms: BHV-7000 75 mg
Drug: Placebo — Matching placebo taken once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether BHV-7000 is effective in the treatment of idiopathic generalized epilepsy with generalized tonic-clonic seizures and includes an additional open-label extension (OLE) phase.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants 18 to 75 years of age at time of consent.
* Diagnosis of Idiopathic Generalized Epilepsy at least 6 months prior to the screening visit, defined by 2017 International League Against Epilepsy (ILAE) Classification and based on requirements of Epilepsy Adjudication criteria.

  1. Subject has probable GTC seizures in the setting of IGE, meaning GTC seizures and either classic 3-4 Hz generalized spike-wave (GSW) or 4-6 Hz polyspike-wave on EEG and no focal abnormality (asymmetric spike-wave fragment is allowed) AND/OR a clear history of absence seizures or myoclonic jerks
  2. Subjects with possible GTC seizures in the setting of IGE, meaning GTC and either Normal EEG OR Generalized epileptiform EEG abnormality with atypical spike-wave and no focal abnormality (asymmetric spike-wave fragment is allowed).
* Subject meets the 2009 ILAE definition of drug resistant epilepsy, failure of adequate trials of two tolerated and appropriately chosen and used ASM schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom.
* Ability of subject or caregiver to keep accurate seizure diaries
* Current treatment with at least 1 to 3 ASMs as part of no more than 4 epilepsy treatments in total (e.g., each ASM is considered 1 treatment. Other epilepsy therapies including devices and diet therapy are allowed; together these other therapies count as 1 treatment).
* Accurate history of having at least 3 days with a GTC seizure evenly spread throughout the 16 weeks prior to the screening visit, such that a subject had at least 1 day with a GTC seizure during the first 8 weeks and at least 1 day with a GTC seizure during the second 8 weeks.

Exclusion Criteria:

* History of status epilepticus (convulsive status epilepticus for > 5 minutes or focal status epilepticus with impaired conscious for > 10 minutes) within the last 6 months prior to screening visit that is not consistent with the subject's habitual seizure.
* History of repetitive/cluster GTC seizures (where individual seizures cannot be counted) within the last 6 months prior to screening visit, or having repetitive/cluster GTC seizures count during the screening phase.
* Any condition that would interfere with and/or confound the interpretation of safety or efficacy data from the study, as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time to the Second Day with a Generalized Tonic Clonic (GTC) Seizure During the 24- week Double-blind Treatment Period | Baseline to Week 24 of Double-Blind Treatment Period
  To compare the efficacy of BHV-7000 to placebo as adjunctive therapy for subjects with idiopathic generalized epilepsy with generalized tonic-clonic (GTC) seizures as measured by the time to the second day with a GTC seizure during the double-blind phase

SECONDARY OUTCOMES:
Percentage of Participants with freedom of GTC seizures during DBT Phase | Baseline to Week 24 of Double-Blind Treatment Period
  To compare the efficacy of BHV-7000 to placebo in terms of the proportion of subjects that are free of GTC seizures as measured by the proportion of subjects with GTC seizure freedom during the 24-week DBP, estimated using Kaplan- Meier methods.
Number of Participants With Deaths, Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and moderate or severe AEs | Baseline to Week 24 of Double-Blind Treatment Period
  To assess the safety and tolerability of BHV-7000 as measured by the number of unique subjects with deaths, SAEs, AEs leading to discontinuation, and moderate and severe AEs
Number of Participants With Clinically Significant Laboratory Abnormalities | Baseline to Week 24 of Double-Blind Treatment Period
  To assess the safety and tolerability of BHV-7000 as measured by the number of unique subjects with grade 3 and grade 4 laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (109):
- United States (40):
  - Accel Research, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - ARENSIA Exploratory Medicine, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Profound Research LLC, Pasadena, California
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - Nova Clinical Research, LLC, Bradenton, Florida
  - University of Florida (Jacksonville), Jacksonville, Florida
  - Y&L Advance Health Care,Inc d/b/a Elite Clinical Research, Miami, Florida
  - Serenity Research Center, Miami, Florida
  - Research Institute of Orlando, Orlando, Florida
  - Comprehensive Neurology Clinic, Orlando, Florida
  - Knight Neurology, Rockledge, Florida
  - Santos Research Center, Tampa, Florida
  - Encore Medical Research of Weston LLC., Weston, Florida
  - Augusta University, Augusta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants in Epilepsy & Neurology, PLLC (CEN), Boise, Idaho
  - Northwestern Medical Group, Department of Neurology, Chicago, Illinois
  - Revive Research Institute, Inc., Elgin, Illinois
  - Bluegrass Epilepsy Research, Lexington, Kentucky
  - OLOLRMC, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Somnos Clinical Research, Lincoln, Nebraska
  - NEREG, Hackensack, New Jersey
  - Institute of Neurology and Neurosurgery, Livingston, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - Boston Children's Health Physicians (BCHP), Hawthorne, New York
  - Northwell Health Pediatric Neurology, New Hyde Park, New York
  - NYU Langone Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - UPMC, Pittsburgh, Pennsylvania
  - WR-ClinSearch, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - ANESC Research, El Paso, Texas
  - Road Runner Research, Ltd, San Antonio, Texas
  - Intermountain Health, Murray, Utah
  - Henrico Doctors' Neurology Associates, LLC, Richmond, Virginia
- Australia (6):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - St Vincents Hospital Melbourne - PPDS, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Christian Doppler-Klinik - Universitätsklinikum der PMU, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - CHU UCL Namur - Site Godinne, Yvoir, Namur
  - UZ Gent, Ghent, Oost-Vlaanderen
- Croatia (2):
  - Clinical Hospital Dubrava, Zagreb, City of Zagreb
  - Clinical Hospital Sveti Duh, Zagreb, City of Zagreb
- Helsinki University Hospital, Helsinki, Uusimaa, Finland
- France (6):
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg, Bas-Rhin
  - CHU Dijon Bourgogne, Dijon, Côte-d'Or
  - CHU de Toulouse-Hôpital Pierre-Paul Riquet-Site de Purpan, Toulouse, Haute-Garonne
  - CHRU Lille, Lille, Nord
  - Hospices Civils de Lyon - 59 Bd Pinel, Bron, Rhône
  - Hôpital Pontchaillou, Rennes
- Germany (11):
  - Epilepsiezentrum Kork, Kehl, Baden-Wurttemberg
  - Universitätsklinikum Ulm-Oberer Eselsberg 45, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - LMU Klinikum der Universität München - Campus Großhadern, München, Bavaria
  - Klinikum der Johann-Wolfgang Goethe-Universitat - Schleusenweg 2-16, Frankfurt am Main, Hesse
  - Universitätsklinikum Gießen und Marburg GmbH - Standort Marburg, Marburg, Hesse
  - Krankenhaus Mara gGmbH, Bielefeld, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Kleinwachau Sächsisches Epilepsiezentrum Radeberg Gemeinnützige Gmbh, Radeberg, Saxony
  - Vivantes - Humboldt Klinikum, Berlin
  - Epilepsie-Zentrum Bodensee, Ravensburg
- Italy (14):
  - Ospedale Policlinico SS Annunziata - Chieti, Chieti, Abruzzo
  - Azienda Ospedaliera Universitaria Renato Dulbecco - AO Mater Domini, Catanzaro, Calabria
  - AORN Antonio Cardarelli, Napoli, Campania
  - AUSL di Bologna - Ospedale Bellaria, Bologna, Emilia-Romagna
  - IRCCS Istituto Neurologico Mediterraneo Neuromed, Pozzilli, Isernia
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - IRCCS Ospedale Pediatrico Bambino Gesù - INCIPIT - PIN, Rome, Lazio
  - Istituto G Gaslini Ospedale Pediatrico IRCCS - INCIPIT - PIN, Genoa, Liguria
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - ASST Santi Paolo e Carlo - Azienda Universitaria-Polo Universitario San Paolo, Milan, Lombardy
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino IRCCS, Pavia, Lombardy
  - Azienda Ospedaliero-Universitaria di Modena - Ospedale Civile di Baggiovara, Baggiovara, Modena
  - Fondazione Policlinico Universitario A Gemelli - Rome - PPDS, Roma
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona
- Kempenhaeghe - PPDS, Heeze, North Brabant, Netherlands
- Poland (6):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Pratia MCM KrakÛw, Krakow, Lesser Poland Voivodeship
  - Twoja Przychodnia-Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - Santa Familia PTG Lodz, Lódz, Lódzkie
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Neurosphera SP. Z O.O Warsaw, Warsaw
- Portugal (5):
  - ULS de Entre Douro e Vouga, EPE - Hospital de São Sebastião, Santa Maria da Feira, Aveiro District
  - ULS de Matosinhos, EPE - Hospital Pedro Hispano, Senhora da Hora, Porto District
  - Centro Clínico Académico, Braga - Hospital de Braga, Braga
  - ULS de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - Hospital da Luz Torres de Lisboa, Lisbon
- Spain (7):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital del Mar, Barcelona
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Centro de Neurologia Avanzada, Seville
  - Hospital Clinico Universitario de Valladolid, Valladolid
- United Kingdom (5):
  - Neuroscience Research Centre, Fazakerley
  - University College London Hospitals, London
  - Morriston Hospital, Morriston
  - The Royal Victoria Infirmary, Newcastle upon Tyne
  - Salford Royal Hospital, Salford